CLINICAL TRIAL: NCT01803815
Title: Evaluation of Antihypertensive Drugs in Patients With Obstructive Sleep Apnea
Brief Title: Evaluation of Antihypertensive Drugs in OSA Patients
Acronym: ADOSA
Status: Completed | Type: Observational
Sponsor: Universidade Nova de Lisboa (Other)
Responsible Party: Sponsor
Other Study IDs: NOVA - CEDOC/FCT
Record Dates: First submitted 2013-02-27; First posted 2013-03-04 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Hypertension; Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; hypertension; antihypertensive drugs
MeSH Terms: conditions — Hypertension; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This prospective cohort study aimed to assess the phenotypic characteristics of OSA patients and their pattern of antihypertensive drugs consumption. The investigators also aimed to investigate a hypothetical association between ongoing anti-hypertensive regimen and Blood pressure control rates in these patients. Additionally, the investigators were also interested in trying to understand if the control of OSA may be influenced by the use of different classes of anti-hypertensive drugs.

ELIGIBILITY:
Inclusion Criteria:

* aged above 18 years, that attended a first visit at CHLN Hospital Sleep Unit were enrolled

Exclusion Criteria:

* severe psychiatric disease or inability to understand the information required for an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients, male and women, aged above 18 years, that attended a first visit at CHLN Hospital Sleep Unit, located in Lisbon, were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2010-04; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with uncontrolled BP before CPAP (Continuous Positive Airway Pressure) adaptation. | patients will be followed up for an expected average time of 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Lucilia N Diogo, PharmD, MSc, Principal Investigator — Universidade Nova de Lisboa - CEDOC; Paula Pinto, PhD, MD, Study Chair — CHLN; Cristina Bárbara, PhD, MD, Study Chair — CHLN; Emilia C Monteiro, PhD, MD, Study Director — Universidade Nova de Lisboa; Ana L Papoila, PhD, Study Director — Universidade Nova de Lisboa
Locations (1):
- Universidade Nova de Lisboa - Faculdade de Ciências Médicas, Lisbon, Portugal